CLINICAL TRIAL: NCT04017767
Title: Intermittent Hypoxia (IH), Respiratory and Motor Plasticity, and Sleep Apnea in Spinal Cord Injury (SCI)
Brief Title: Motor Plasticity, Intermittent Hypoxia and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Shirin Shafazand, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20190415
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea, Obstructive; Spinal Cord Injuries; Hypoxia
Keywords: Neuroplasticity; Respiratory Function; Motor Function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Spinal Cord Injuries; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: subjects with OSA compared to subjects without OSA based on their response to IH (intermittent hypoxia) exposure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate to Severe Obstructive Sleep Apnea (OSA) (Experimental): Individuals with moderate to severe OSA defined as having an Apnea-hypopnea Index (AHI) that is greater than or equal to 15.
  Interventions: Procedure: Induced Acute Intermittent Hypoxia (AIH); Device: AIH mask
- Without OSA (Active Comparator): Individuals without OSA defined as having AHI less than 5.
  Interventions: Procedure: Induced Acute Intermittent Hypoxia (AIH); Device: AIH mask

INTERVENTIONS:
Procedure: Induced Acute Intermittent Hypoxia (AIH) — AIH will be administered on days 1-3. Each day entails 15 and 90 second hypoxic intervals (Fraction of Inspired Oxygen (FIO2) = 0.09) alternating with 60-second normoxic intervals (FIO2 = 0.21).
Device: AIH mask — Induced Intermitted hypoxia will be delivered via the AIH mask. The mask has two one-way valves restricting inspiration to the top valve and expiration to the bottom valve. Hypoxic and normoxic gas mixtures will be delivered through the top valve.

SUMMARY:
The purpose of this study is to learn about the effect of sleep apnea and low oxygen on muscle strength and lung function in people with chronic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older,
2. Chronic (≥ 1-year post-injury), non-progressive SCI,
3. Asia Impairment Scale (AIS) C or D,
4. Resting Saturated oxygen (SaO2) ≥ 95%,
5. Cervical injury (C5-C8)

Exclusion Criteria:

1. Currently hospitalized,
2. Resting heart rate ≥120 Beats per minute (BPM),
3. Resting systolic blood pressure >180 mmHg,
4. Resting diastolic Blood Pressure >100 mmHg,
5. Self-reported history of unstable angina or myocardial infarction within the previous month,
6. OSA that is being treated with positive airway pressure therapy,
7. Women who know or suspect they may be pregnant or who may become pregnant,
8. Known underlying lung disease,
9. Pregnant Women,
10. Prisoners,
11. Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The difference in Motor Function assessed via hand grip strength measured by maximum grip strength (MGS) between participants with moderate to severe OSA and without OSA. | Baseline
  Participants will be instructed to squeeze the hand grip dynamometer with maximal effort for 3-5 seconds. This will be repeated three times for each hand with 1 minute of rest between trials. The highest value obtained will be used as the MGS.
The difference in Motor Function assessed via hand grip strength measured by electromyographic (EMG) recordings between participants with moderate to severe OSA and without OSA. | Baseline
  Electrodes will be secured on the participant to measure EMG. Participants will then be asked to press the index finger against a custom lever. The participant will perform three brief maximal voluntary contractions (MVC) for 3-5 seconds separated by 60 seconds of rest. The highest of the three values will be used.

SECONDARY OUTCOMES:
Change in Motor Function assessed via hand grip strength measured by MGS. | Baseline to Day 1 post AIH, Baseline to Day 3 post AIH, Baseline to Day 10, Baseline to Day 17
  Participants will be instructed to squeeze the hand grip dynamometer with maximal effort for 3-5 seconds. This will be repeated three times for each hand with 1 minute of rest between trials. The highest value obtained will be used as the MGS.
Change in Motor Function assessed via hand grip strength measured by EMG recordings. | Baseline to Day 1 post AIH, Baseline to Day 3 post AIH, Baseline to Day 10, Baseline to Day 17
  Electrodes will be secured on the participant to measure EMG. Participants will then be asked to press the index finger against a custom lever. The participant will perform three brief maximal voluntary contractions (MVC) for 3-5 seconds separated by 60 seconds of rest. The highest of the three values will be used.
Change in biomarker levels | Baseline to Day 1 post AIH, Baseline to Day 3 post AIH, Baseline to Day 10, Baseline to Day 17
  Serum Brain-Derived Neurotrophic Factor (BDNF) and Vascular Endothelial Growth Factor (VEGF) biomarker levels in pg/ml will be evaluated. At baseline, the blood samples will be collected after 12 hours of overnight fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Shafazand, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No